CLINICAL TRIAL: NCT02990546
Title: Midodrine Use in the Recovery Phase of Septic Shock
Brief Title: Midodrine in the Recovery Phase of Septic Shock
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Unable to enroll subjects before PI left institution
Sponsor: University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19198
Record Dates: First submitted 2016-11-16; First posted 2016-12-13 (Estimated); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Midodrine; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): In the intervention arm 10 mg of midodrine will be given orally three times daily starting at the time of stable or decreasing intravenous vasopressor support
  Interventions: Drug: midodrine
- Control (Other): The control arm will receive standard of care for septic shock with IV vasopressor support as needed to maintain MAP goal > 65 mmHg
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: midodrine — Midodrine will be given to treatment arm as enteral medication
  Other Names: Midodrine Hydrochloride; Proamatine
  Arms: Intervention
Other: Standard of Care — Patients in the control arm will receive standard of care for septic shock
  Arms: Control

SUMMARY:
The aim of this study is to investigate the role of oral midodrine in the recovery of septic shock. The investigators hypothesize that the oral drug can reduce central line days and ICU length of stay.

DETAILED DESCRIPTION:
The investigators aim to investigate the use of midodrine in the recovery phase of septic shock in a randomized control trial. The investigators hypothesize that midodrine use initiated after stabilization or improving intravenous vasopressor requirement will lead to decreased length of ICU stay and length of time that intravenous vasopressors are required.

The investigators plan to enroll and consent patients at the onset of septic shock. Once IV vasopressor requirement is stabilized or decreasing, males and females will be randomized in 1:1 fashion to receive either standard clinical care or standard clinical care plus oral midodrine. The investigators will analyze length of stay in the ICU, time on vasopressors, time needing a central line, and hospital length of stay.

ELIGIBILITY:
Inclusion Criteria:

* • Patients aged 18-99 years old

  * Admitted to UVA medical ICU with diagnosis of septic shock.

Exclusion Criteria:

* Pregnant females, patients with childbearing potential will have urine pregnancy testing after consent
* Patients < 18 years
* Prisoners
* Patients already taking midodrine
* Patients with cirrhosis and Child-Pugh Class C (Child-Pugh score > 9)_
* Patients with Increased intraocular pressure and glaucoma
* Patients with allergy to midodrine
* Non-English speaking patients
* Patients without enteral access
* Patients where the attending physician does not feel MAP goal of > 65 mmHg is physiologically acceptable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-02 (Actual)

PRIMARY OUTCOMES:
ICU free days | 28 days
  ICU free days from first 28 days

SECONDARY OUTCOMES:
Central venous catheter free days | 28 days
IV vasopressor free days | 28 days
Hospital length of stay | up to 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Jones, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No